CLINICAL TRIAL: NCT01732133
Title: Evaluation of the System NEXFIN for Continuous and Non-invasive Measure of the Blood Pressure During Cesarean Delivery Practised Under Spinal Anesthesia
Brief Title: Evaluation of NEXFIN During Cesarean Delivery to Detect Hypotension
Acronym: NEXFIN-CESAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/27; 2012-A00811-42 (Other: ANSM)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Hypotension
Keywords: Hypotension; Cesarean delivery
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Measurement of arterial pressure (Experimental)
  Interventions: Device: Nexfin

INTERVENTIONS:
Device: Nexfin
  Other Names: Continuous measurement of arterial pressure using Nexfin

SUMMARY:
Hypotension after spinal anesthesia for cesarean delivery occurs frequently. Oscillometric measurement gives intermittent informations. Nexfin, a continuous noninvasive device, could help to detect hypotension.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing elective cesarean delivery performed under spinal anesthesia

Exclusion Criteria:

* patients with a heart rhythm disorder, Raynaud's disease or a history of vascular surgery of the upper limb

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-01-22 (Actual); Study Completion 2016-01-22 (Actual)

PRIMARY OUTCOMES:
Comparison between Nexfin and intermittent measurements of blood pressure | two years
  Bland and Altman analysis (bias and limits of agreement). Analysis concerns data from intrathecal injection to childbirth

SECONDARY OUTCOMES:
Area under the curve between both measurements | two years
  Analysis concerns data from intrathecal injection to childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch
Locations (2):
- France (2):
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Hopital Foch, Suresnes

REFERENCES:
- [Derived] Bobet M, Joachim J, Gayat E, Bonnet A, Sievert K, Barnichon C, Fischler M, Le Guen M. Blood pressure measurement during cesarean delivery: Evaluation of a beat-to-beat noninvasive device (NexfinTM). Medicine (Baltimore). 2021 Jun 4;100(22):e26129. doi: 10.1097/MD.0000000000026129. PMID 34087863